CLINICAL TRIAL: NCT02113904
Title: Phase II Clinical Trial Using Humira in Netherton Syndrome
Brief Title: Clinical Trial Using Humira in Netherton Syndrome
Acronym: AntiTNF-SN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P100150; 2013-002205-54 (EudraCT Number)
Record Dates: First submitted 2014-04-02; First posted 2014-04-15 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Netherton Syndrome
Keywords: Netherton syndrome; Adalimumab; TNF-alpha; Orphan genetic syndrome
MeSH Terms: conditions — Netherton Syndrome | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adalimumab (Experimental)
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — 6 injections (one every 15 days during 3 months)
  Other Names: Humira

SUMMARY:
The main objective of this studies therapeutic : to determine the effect of Adalimumab (HumiraR) on clinical inflammatory manifestations of patients with Netherton syndrome after 3 months of treatment , with a post treatment period follow-up of 3 months.

Second objectives are To evaluate the safety of Adalimumab in the context of NS To evaluate the improvement of the quality of life at 3 months To evaluate the improvement of pruritus and pain in the patients To study markers of inflammatory and allergy in NS prior and after treatment Benefit of the study An improvement by at least 20% of the cutaneous signs in these patients who suffer from a genetic incurable, chronic, painful and very afflicting disease would be of a great help for these patients. NS is a major source of social exclusion.

Risks They are inherent to the risks of biotherapies, especially for an anti-TNF therapy, they comprise a risk of infection. Cutaneous infections occur mainly during infancy, and we have therefore chosen to treat patients over 4 years of age in this study.

A close clinical surveillance will be set up (initially every week during the first month of treatment, then every month). This will represents a large number of visits but will provide a high level of security.

Benefits/risks ratio In the absence of curative treatment for these patients with a severe genetic skin disease, the benefits/risks ration clearly appears to be in favour of an expected benefit.

DETAILED DESCRIPTION:
Netherton syndrome (NS) is a rare (incidence is estimated at 1 in 100 000) but severe genetic skin disease characterized by scaly erythroderma at birth, abnormal hair and severe psoriasiform /atopic dermatitis-like lesions with high IgE levels and allergic manifestations. It has considerable impact on the quality of life of patients, as a result of inflammatory and painful flares, the chronicity of the lesions, severe growth retardation with definitive short stature.

NS is caused by loss of function SPINK5 mutations which lead to unregulated epidermal protease activity : kallikrein 5, kallikrein 7 and elastase proteases are found overactive following loss of inhibition. Secondly, KLK5 activates PAR-2 receptors at the keratinocyte surface leading to the activation of the NF-KB pathway and the release of different pro-inflammatory cytokines such TNF-alpha .

There is no specific treatment for NS. The different therapeutic attempts by Soriatane (acitretin) have worsen the skin inflammation and dryness. The use of topical calcineurin inhibitors (Tacrolimus) has sometimes improved skin inflammation but with an important systemic diffusion. The use of immune suppressive drugs in severe patients with NS followed in our labelized Centre (Cyclosporine, methotrexate, mycophenolate mofetil) have not brought a significant and durable improvement. So NS is a very distressing genodermatosis.

For these clinical and biological considerations, a benefit with anti TNF treatment could be expected and the evaluation of such treatment is justified in NS. The clinical case of an adult patient with severe NS, improved by anti-Tnf treatment has recently been published in the literature

ELIGIBILITY:
Inclusion Criteria:

* Patient over 4 years of age at the time of enrolment
* Patient with a clinical, immuno-histochemical and/or molecular diagnosis confirmed
* Vaccinations to date
* Informed consent form signed by the patient and/or his parents (or the legal authority) if the patient is a child
* Patient with social security coverage

Exclusion Criteria:

* Ongoing severe infections
* Well known allergy to one of Adalimumab ingredients
* Allergy to xylocaine
* Ongoing treatment to immunosuppressive drugs and biotherapies
* History of malignancy
* Heart, renal, haematological and/or confirmed hepatic involvement
* Pregnant, or breastfeeding, patients
* Anomalies of the standard balance sheet: neutropenia < 1000/mm3, polynucleose > 12 000 / mm3 - lymphopenia < 1000 / mm3 - anemia < 9g / 100ml - thrombocytopenia < 150 000 /mm3, thrombocytosis > 500 000/mm3 - transaminase > 3N

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-01-27 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
SN-EASI score and EASI score | month 3
  To evaluate the severity of specific netherthon syndrome clinical manifestation and the severity of atopic dermatitis before treatment, after three months of treatment, after a period of three months without treatment

SECONDARY OUTCOMES:
SN-EASI score and EASI score | at inclusion before treatment
  To evaluate the severity of specific netherthon syndrome clinical manifestation and the severity of atopic dermatitis before treatment, after three months of treatment, after a period of three months without treatment
SN-EASI score and EASI score | month 6
  To evaluate the severity of specific netherthon syndrome clinical manifestation and the severity of atopic dermatitis before treatment, after three months of treatment, after a period of three months without treatment
Number of participants with adverse events | month 3
  To evaluate the safety of adalimumab for netherton syndrome patients
CDLQI and DLQI | at inclusion before treatment
  To evaluate the quality of life of the patients
CDLQI and DLQI | month 3
  To evaluate the quality of life of the patients
CDLQI and DLQI | month 6
  To evaluate the quality of life of the patients
Improvement of pain | month 3
  Visual scale from 0 to 10
Improvement of pruritus | month 3
  Visual scale from 0 to 10
Hair growth | month 3
  Visual scale from 1 to 4
Circulating inflammatory response (pro-inflammatory cytokines) cutaneous inflammatory response | month 3
  Markers of inflammatory response before and after treatment
Circulating inflammatory response (pro-inflammatory cytokines) cutaneous inflammatory response | month 6
  Markers of inflammatory response before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christine Bodemer, MD, PhD, Study Chair — : Department of Dermatology, Necker Enfants malades hospital, University Paris Descartes 149 rue de sèvres 75015 Paris, France
Locations (1):
- Necker Enfants Malades hospital, Paris, France